CLINICAL TRIAL: NCT02025140
Title: Comparison of The Computer Controlled Local Anesthesia and The Conventional Inferior Alveolar Nerve Block in Primary Molars Pulptomies
Brief Title: Computer Controlled Local Anesthesia in Children
Acronym: STA machine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, DR.Khlood Baghlaf, DR, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2013-11-25; First posted 2013-12-31 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Pain Perception of the New Device; The Pain Related Behavior; The Effectiveness of Anesthesia
Keywords: Computer controlled anesthesia (CCLAD); pain perception; Effectiveness; primary molars; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- : This group consisted of 30 patients. (Active Comparator): The traditional IANB injection was given according to the standard technique (Evers and Haegerstam 1981). From everyday practice, it is known that the present operator takes approximately 60 to 90 seconds to give a mandibular block
  Interventions: Device: conventional anesthesia syringe
- 30 IANB with Computer controlled (Experimental): The IANB injection was given by a computer- regulated device performed with the STA system. The IANB injection was given according to the manufacturer's instruction (the model was used is the STA Single Tooth Anesthesia System produced by Milestone Scientific, Livingston, NJ).
  Interventions: Device: Computer controlled anesthesia
- consisted of 30 periodontal anesthesia (Experimental): The interligamental injection was given by computer- regulated device performed with the STA system.
  Interventions: Device: Computer controlled anesthesia

INTERVENTIONS:
Device: Computer controlled anesthesia — The IANB by the computer controlled local anesthetic device CCLAD and periodontal ligament anesthesia by the CCLAD
  Other Names: (The Wand); STA machine
  Arms: 30 IANB with Computer controlled; consisted of 30 periodontal anesthesia
Device: conventional anesthesia syringe — Active control
  Other Names: Inferior alveolar nerve block injection
  Arms: : This group consisted of 30 patients.

SUMMARY:
• Introduction: Effective pain control is critical in pediatric dentistry. The effectiveness of pain control in children can be influenced by child characteristics .

Objectives: The Purpose of the study is to compare the pain perception and the effectiveness of anesthesia between the computer-controlled local anesthetic delivery system (CCLAD) and the traditional inferior alveolar nerve block (IANB) in pulptomies of the mandibular second primary molars.

Materials and Methodology: The study sample includes 90 healthy children who are selected randomly from the R4 electronic filing system in King Abdulaziz University Hospital (KAUH) with age range from 5-9 years. The child is required local anesthesia for pulpotomies in the mandibular second molars. The sample will be divided randomly to one of these 3 groups: group A is composed of 30 patients who will be anesthetized by the traditional IANB. Group B includes 30 patients will be anesthetized by the IANB using CCLAD. While, the remaining 30 patients will be assigned in group C and will be anesthetized by periodontal ligament injection anesthesia using the CCLAD. The pain perception levels after the injection is assessed by a Wing-Baker faces pain scale. Effectiveness of the anesthesia during each step in pulpotomy is measured using Sounds, eyes and motor (SEM) scale. After the treatment by 24 hours parents will be contacted by the telephone to ask about the presence of postoperative pain or lip biting. Statistical analysis is carried out using SPSS version 16.00.

DETAILED DESCRIPTION:
Ethical Consideration:

The Ethical Committee of King Abdulaziz University KAAUEC approved the study .

Subjects' selection:

The Sample includes children who are randomly selected by the R4 electronic file system in the pediatric dentistry specialty clinics at King Abdulaziz University Hospital (KAUH). A total of 2100 pediatric screening had been registered between April 2013 and November 2013 .These files will be checked for the eligible age in the study which is 5-9 years. Then, the inclusion and exclusion criteria will be checked, and the patients will be selected by systemic random sample.

Study design:

This is a randomized single blind clinical trial study.

ELIGIBILITY:
The inclusion criteria:

1. Age of the children was ranged from 5-9 years.
2. Children were healthy physically and mentally; all children had no contraindications to local anesthesia.
3. Children were assessed as being cooperative, had behavioral ratings "positive" or "definitely positive" according to the Frankl (Frankl et al 1962) behavior classification scale (appendix1).
4. Children were diagnosed with carious mandibular second primary molars that required treatment with pulpotomies.

The exclusion criteria:

1. Disapproved consent.
2. Medically compromised children.
3. Uncooperative children.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The pain perception of the children to the device | 1-2 minutes
  No follow up is required, the out come is measured immediately after completion of the injection

SECONDARY OUTCOMES:
The effectiveness of the anesthesia | During the procedure
  The sound eye motor scale is used during different stages of procedure.

OTHER OUTCOMES:
The pain related behavior | 1-2 minutes
  The established behavior code was used during administration of the injection

CONTACTS AND LOCATIONS:
Overall Officials: Prof Najlaa M Alamoudi, PHD, Principal Investigator — King Abdulazize University
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

REFERENCES:
- See also: Related Info — http://www.milestonescientific.com/dental